CLINICAL TRIAL: NCT02127723
Title: An Open, Non-comparative Single Center Study to Evaluate Efficacy and Safety of HA (Macrolane VR30) in Buttocks Reshaping and Contouring
Brief Title: (Macrolane VR30) in Buttocks Reshaping and contouringCellulite (Macrolane VR30) in Buttocks Reshaping and Contouring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31GC1202
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2020-09

CONDITIONS: Cellulite of the Buttocks
Keywords: cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macrolane (Experimental): All subjects will receive hyaluronic acid injection (Macrolane VRF30)
  Interventions: Device: Hyaluronic acid injection (Macrolane VRF30)

INTERVENTIONS:
Device: Hyaluronic acid injection (Macrolane VRF30) — Injection of Macrolane subcutaneously in the buttocks area to reduce cellulite

SUMMARY:
The most common treatments today for enhancing the shape and size of the buttocks are transplantation of the patient's own body fat after liposuction and insertion of permanent implants. Macrolane VRF30 is a gel product based on hyaluronic acid which is a transparent slow-flowing gel. A similar hyaluronic-acid gel from the same manufacturer, Q-Med AB, has been used for many years for the treatment of facial wrinkles. By injecting Macrolane gel into the skin, the shape of the buttocks can be altered and their volume increased.

DETAILED DESCRIPTION:
Aesthetic dermatologists have reported promising results on the use of Macrolane VRF30 for buttocks reshaping and contouring. Although treatment with Macrolane VRF is well documented in breast enhancement, there is limited documentation on the use in buttocks reshaping. Based on these clinical impressions, this study aims at acquiring information on the efficacy and safety of Macrolane VRF30 in this particular indication. As a result of the reshaping of the buttocks, it is expected that improvement of skin laxity will result in contouring and reduction of cellulite. By using standardised evaluation tools, the results of buttock reshaping reported anecdotally can be confirmed by accurate measurements.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female subjects older than 30 years. 2. Subjects presenting with loss of contour of the upper half of the buttocks, associated with skin laxity and appearance of cellulite grade 1 or 2 on items A, B and D of the CSS.

  3. Treatment-naïve subjects for fillers in the areas to be treated. 4. Subjects with signed informed consent. 5. Medical history and physical examination which, based on the investigator's opinion, do not prevent the subject from taking part in the study and use the product under investigation.

  6. Subjects should maintain their habits regarding physical activity. 7. Availability of the subject throughout the duration of the study.

Exclusion Criteria:

* 1. Pregnant women or women intending to get pregnant in the next 12 months. 2. Subjects with known hypersensitivity to any compound of the study product or anaesthesia used in the study.

  3. Subjects with history of any other adverse effect, which should prevent the subject from participating in the study according to the investigator's opinion.

  4. Subjects participating in other clinical trials within 30 days prior to baseline.

  5. Any prior surgery, any prior cosmetic procedures or side effects from previous procedures in the buttocks, including permanent fillers, liposuction and prosthesis, that may interfere with the results.

  6. Subjects with presence of autoimmune disease or other chronic disease that in the opinion of the Investigator may interfere with the outcome of the study.

  7. Subjects on immunomodulatory therapy (suppressive or stimulatory). 8. Subjects with active inflammation or infection in the areas to be treated. 9. Subject with bleeding disorders or subjects who are taking thrombolytics or anticoagulants.

  10. Subjects who have taken inhibitors of platelet aggregation, including nonsteroidal anti-inflammatory agents and acetylsalicylic acid, 2 weeks before treatment.

  11. Subjects with contraindications for MRI, such as presence of pacemaker, clips or splinter, metal prosthesis or tendency for claustrophobia.

  12. Subjects who are study site staff for this study, or close relatives of the study site staff, as well as subjects who are employed by the Sponsor company, or close relatives of employees at the Sponsor company.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris Hexsel, Dr, Principal Investigator — Brazilian Center for Studies in Dermatology
Locations (1):
- Dr Hexsel, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Macrolane: All subjects will be treated with Macrolane
  Hyaluronic acid injection (Macrolane VRF30): Injection of Macrolane subcutaneously in the buttocks area to reduce cellulite
Period: Overall Study
Arm/Group | Macrolane
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Macrolane: Att subjects will be treated with Macrolane
  Hyaluronic acid injection (Macrolane VRF30): Injection of Macrolane subcutaneously in the buttocks area to reduce cellulite
Arm/Group | Macrolane
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 20
Cellulite severity scale [Mean (Standard Deviation); unit: units on a scale] — A scale graded 1-15 that measures the severity of cellulites. Grade 1-5 is mild; grade 6-10 is moderate; grade 11-15 is severe.
  units on a scale | 8 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Aesthetic Improvement of the Buttocks Using Investigator GAIS
Description: Assess the aesthetic improvement of the buttocks after reshaping in female subjects with cellulite associated with laxity and loss of volume of the buttocks at each follow up visit after treatment using the investigator Global Aesthetic Improvement Scale (GAIS).
Time Frame: 48 weeks post treatment
Population: Global aesthetic improvement was assessed as Very much improved, Much improved, Improved, No change or Worse. Number of improved subjects (i.e. very much improved, much improved or improved) was presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Macrolane
Number analyzed (Participants) | 19
Participants | 7

2. Primary Outcome: Mean Improvement in Cellulite Severity Compared to Baseline Using the Cellulite Severity Scale (CSS)
Description: Assess improvement of cellulite in the buttock areas compared to baseline at each follow up visit after treatment using the Cellulite Severity Scale (CSS). A scale graded 1-15 that measures the severity of cellulites. Grade 1-5 is mild; grade 6-10 is moderate; grade 11-15 is severe.
Time Frame: 48 weeks post treatment
Population: Improvement in cellulite at 48 weeks compared to baseline, using the CSS and indicated by the grading reduction.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Macrolane
Number analyzed (Participants) | 19
Units on a scale | -1 (1.6)

3. Primary Outcome: Number of CSS Responders
Description: Assess the CSS responder rate, where a responder is defined as a subject who has improved at least one grade from baseline in items A and/or B and/or D of the CSS.
Time Frame: 48 weeks post treatment
Population: Number of subjects who were improved at least 1 grade from baseline in items A and/or B and /or D of the CSS.
Measure: Count of Participants; unit: Participants
Arm/Group | Macrolane
Number analyzed (Participants) | 19
Participants | 10

4. Secondary Outcome: Number of Subjects With Related Adverse Events
Description: Number of subjects with related adverse events
Time Frame: Until 48 weeks post treatment
Population: Evaluation of safety by assessment of number of related adverse events (AEs)
Measure: Number; unit: subjects
Arm/Group | Macrolane
Number analyzed (Participants) | 20
subjects | 10

ADVERSE EVENTS:
Arm/Group | Macrolane
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macrolane (N=20)
injection site pain (General disorders) | 8 (14)
injection site hematoma (General disorders) | 2 (3)
injection site puritus (General disorders) | 1 (1)
injection site discomfort (General disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less